CLINICAL TRIAL: NCT05822596
Title: The Effectiveness and Feasibility of Tablet-based Interactive Games in Elderly With Cognitive Impairment and Persons With Intellectual Disability: A Randomised Controlled Trial
Brief Title: Tablet-based Interactive Games in Elderly With Cognitive Impairment and Persons With Intellectual Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tablet games_protocol_v1
Record Dates: First submitted 2023-04-04; First posted 2023-04-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Technology; Cognitive Impairments; Intellectual Disability
Keywords: Gerontechnology; Interactive games; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction; Intellectual Disability

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated into either intervention group and control group in a 1:1 allocation ratio. The target participants are residents in elderly residential settings, members in day care units for the elderly, and persons with intellectual disabilities in day activity centre cum hostel. Participants in the experimental group will participate in a 12-week cognitive training program that includes facilitated sessions and non-facilitated sessions.
Who Masked: Outcomes Assessor
Masking Description: Assessors of the outcomes will not be involved in the recruitment and intervention delivery and will be blinded to group allocation (single blindness).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet-based interactive games experimental group (Experimental): The experimental group will take part in a 12-week cognitive training program using tablet-based interactive games.
  Interventions: Device: Tablet-based interactive games experimental group intervention
- Control group (No Intervention): The control group will receive treatment as usual during the 12-week trial.

INTERVENTIONS:
Device: Tablet-based interactive games experimental group intervention — The program consists of 24 facilitated sessions and, depending on the capability of the participants, the availability of mobile devices and the service setting, 0 - 84 non-facilitated sessions.
  In 30-minute facilitated session, a program facilitator will lead 1-8 participants in playing the tablet-based interactive games and helpers (e.g., health workers, program workers, and volunteers) will assist the program facilitator in running the sessions. The games may be played individually or together with other participants. In non-facilitated sessions, the participants can play cognitive games depending on the capability of themselves and at their own pace for 10 - 30 minutes
  Arms: Tablet-based interactive games experimental group

SUMMARY:
The study has 10 research questions regarding the cognitive training program and tablet-based interactive games:

Primary study questions:

1. Can the participation of 12-week cognitive training program using tablet-based interactive games maintain cognitive functioning?

   Secondary study questions:
2. Can the participation of 12-week cognitive training program using tablet-based interactive games improve the scores of 6 supplier-developed cognitive domains (including executive function, memory, eye-hand coordination, attention, visual-spatial ability, language)?
3. Can the participation of 12-week cognitive training program using tablet-based interactive games improve the reaction time of the participants?
4. What is the attendance rate in the cognitive training program, and for how long do the participants play the tablet-based interactive games?
5. What is the usability and acceptability of the tablet-based interactive games?

   Auxiliary study questions:
6. Can the participation of 12-week cognitive training program using tablet-based interactive games reduce neuropsychiatric symptoms?
7. Can the participation of 12-week cognitive training program using tablet-based interactive games improve upper-body flexibility?
8. What are the physical side effects of using digital devices in the 12-week cognitive training program?
9. What are the perceived benefits and feasibility of the cognitive training program and tablet-based interactive games?
10. Can the participation of 12-week cognitive training program using tablet-based interactive games improve activities of daily living of persons with intellectual disability?

DETAILED DESCRIPTION:
Study design

The trial is a randomized controlled trial. The participants will be randomly allocated into either intervention group and control group in a 1:1 allocation ratio. The target participants are residents in elderly residential settings, members in day care units, and persons with intellectual disabilities in day activity centre cum hostel. Participants in the experimental group will participate in a 12-week cognitive training program that includes facilitated sessions and non-facilitated sessions. The outcome indicators between joining and not joining the 12-week cognitive training program will be compared. In addition, the compliance of the participants, the perceived benefits and feasibility of the program and games will be assessed.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP) and Declaration of Helsinki.

Procedures

1. Participants' recruitment and consent

   Elderly with Mild Cognitive Impairment (MCI) in the elderly service setting

   Elderly scoring above the cutoff for dementia in Montral Cognitive Assessment - Hong Kong (MoCA - HK) and not receiving a medical diagnosis of dementia or other mentally incapacitating disease will be classified as competent in giving consent and will be invited to give consent.

   Elderly with dementia & Persons in the rehabilitation setting

   For elderly with dementia scoring below the cutoff in MoCA or receiving a diagnosis of mentally incapacitating disease, and persons in the rehabilitation setting, the criteria stated in the Alzheimer Europe Report (2011) will be followed to ensure that they are provided chances to give consent. In particular, four criteria will be evaluated, including 1) the person must have sufficient capacity to understand the information, 2) the person is able to retain, use and weight up such information for making a decision, 3) the person will understand the benefit, risk, and convenience, 4) the person must have the ability to communicate the decision. The University of Hong Kong (HKU) research staff and the care staff will first commit them in a causal chat to assess their ability to communicate and understand the dialogues.

   If potential participants are competent in giving consent, both potential participants and their next of kin members will be approached for consent. In cases potential participants are not competent in giving consents, only their next of kin will be approached for consent. They will then be referred to join a 1-to-1 study introduction session. In this session, HKU research staff and service unit staff will introduce the study to the participant, and invite them to sign a consent form.

   For program facilitators, written consent will be obtained from them before qualitative interviews.
2. Randomization

   After all baseline assessment are completed, participants will be individually randomized to experimental group or control group. A list of random numbers will be generated to create a list of random group allocation (either experimental or control; allocation ratio 1:1), using the RAND function of Excel. The research staff will perform the randomization procedure, by assigning consenting participants who meet all eligibility criteria to the two groups using the list.
3. Training of tablet-based interactive games for program facilitators

   A few identical 60-minute trainings on tablet-based interactive games will be delivered to the program facilitators, who will lead the cognitive training program at the study sites. During the training, they will learn how to operate the game system and lead the participants to play the games. A protocol will be provided for the facilitators in running the program.
4. Pilot run

   The first facilitated and non-facilitated sessions of the 12-week cognitive training program will be used as a pilot run to revise the test protocol and program structure.
5. Implementation

Participants in the experimental group will take part in a 12-week cognitive training program using tablet-based interactive games. The supplier will provide personal accounts to the study sites, so that program facilitators can keep track on the cognitive performance of the individual participant through system reports. Program facilitators will help participants log in the accounts at the start of the facilitated and non-facilitated sessions.

The platform has 79 mini-games that aim to train six cognitive domains, including executive function, memory, eye-hand coordination, attention, visual-spatial ability, and language. Based on the performance and ability of the user, program facilitator can choose the game difficulty level that most fit the participant. To enhance participation, the game utilizes local elements, such as old Hong Kong, supermarkets, and calligraphy. Additionally, some games allow two or more players to participate, for example Mah-jong. During playing the games, the system will assess the cognitive performance of the participants, and calculate a score for each of the six cognitive domains for the program facilitator.

The program consists of 24 facilitated sessions and, depending on the capability of the participants, the availability of mobile devices and the service setting, 0 - 84 non-facilitated sessions.

5.1 Facilitated sessions

There will be two 30-minute facilitated sessions each week. In each session, a program facilitator will lead 1-4 participants in playing the tablet-based interactive games. Helpers (e.g., health workers, program workers, and volunteers) will assist the program facilitator in running the sessions. The games may be played individually or together with other participants.

5.2 Non-facilitated sessions

In non-facilitated sessions, depending on the capability of the participants and the availability of mobile devices, the participants can play cognitive games by themselves and at their own pace for 10 - 30 minutes. In elderly service setting, there will be 0 - 4 non-facilitated sessions per week. In rehabilitation service setting, there will be 0 - 7 non-facilitated sessions per week. These sessions can be administered by staff other than the program facilitators.

5.3 Intervention for control group

During the 12-week trial, the control group will join activities other than the tablet-based interactive games as in experimental group.

To better understand the nature of the control group, the scheduled activities for the control group when the experimental group joins the 12-week training program will be collected.

Blinding

Participants and program facilitators cannot and will not be blinded to the intervention. Assessors of the outcomes will not be involved in the recruitment and intervention delivery and will be blinded to group allocation (single blindness).

Sample size determination

The sample size is estimated by the current number of eligible service users and related staff at the test sites. It is estimated that a total of 81 participants and 10 program facilitators will be recruited.

Data analysis

1. Main analysis

   Linear mixed model analysis will be used to test the interaction between group and time of the outcome indicators of cognitive functioning, reaction time, upper-body flexibility, neuropsychiatric symptoms, activities of daily living, and physical side effects of using digital devices. A partial-eta square will be used to estimate the effect size in comparing the intervention group with the control group. Linear mixed model analysis will also be used to examine the changes in the 6 supplier-developed cognitive domains over time.

   Descriptive statistics will be used to describe the attendance rate in cognitive training program, time spent on playing tablet-based interactive games, and usability and acceptability of the tablet-based interactive games.
2. Qualitative interview

The content will be transcribed verbatim in Chinese for further analysis. Transcripts will be analysed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the tablet-based interactive games. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the service users in elderly service setting:

* Diagnosed with mild to moderate dementia by doctors, or scoring at least 5 and lower than the norm-derived age and education adjusted cutoff scores 7th percentile in HK-MoCA (i.e. elderly with MCI, mild dementia and moderate dementia), and
* Able to understand Chinese

Inclusion criteria for the service users in rehabilitation service setting:

* Aged 40 or above,
* Diagnosed with intellectual disability (IQ<70), and
* Able to understand Chinese

Inclusion criteria for the program facilitators:

* Occupational therapists of the study sites (preferably), or
* Social workers or nurses of the study sites

Exclusion Criteria:

Exclusion criteria for both types of service users:

• Inability to join the intervention program due to severe mental illness, behavior problems, sight impairment, hearing impairment, or communication impairment, as determined by the program facilitator

Exclusion criteria for the program facilitators:

• Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Change of cognitive functioning of elderly without intellectual disability before and after using the tablet-based interactive games | Baseline and at the end of 12-week trial period
  Change of cognitive functioning of elderly without intellectual disability before and after using the tablet-based interactive games will be assessed by HKU research staff who is blinded to group allocation. Total nine items on Hong Kong Brief Cognitive Test (HKBC) will be completed at the baseline and the end of 12-week trial period and the minimum and maximum scores are 0 and 30 respectively.
Change of cognitive functioning of person with intellectual disability before and after using the tablet-based interactive games | Baseline and at the end of 12-week trial period
  Change of cognitive functioning of person with intellectual disability before and after using the tablet-based interactive games will be assessed by HKU research staff who is blinded to the group allocation. Total twenty-one items on 21-item Short Form of the Prudhoe Cognitive Function Test (SF-PCFT) will be completed at the baseline and the end of 12-week trial period and the minimum and maximum scores are 0 and 30 respectively.

SECONDARY OUTCOMES:
The scores of 6 supplier-developed cognitive domains | From the start to the end of 12-week trial period
  The scores of 6 supplier-developed cognitive domains (including executive function, memory, eye-hand coordination, attention, visual-spatial ability, language) in the tablet-based interactive games will be calculated by the game system throughout the program and provided by the supplier.
Change of reaction time before and after using the tablet-based interactive games | Baseline and at the end of 12-week trial period
  Change of reaction time before and after using the tablet-based interactive games will be assessed by HKU research staff who is blinded to the group allocation. Human Benchmark: Reaction time (https://humanbenchmark.com/tests/reactiontime) will be used to assess at the baseline and the end of 12-week trial period. In each assessment, the participants will undergo the test for four trials. The average reaction time in terms of mini-seconds of the trials will be recorded.
Attendance rate in the cognitive training program (including facilitated and non-facilitated sessions) | From the start to the end of 12-week trial period
  Attendance rate in cognitive training program (including facilitated and non-facilitated sessions) will be recorded by the game system and provided by the supplier.
Time spent on playing tablet-based interactive games | From the start to the end of 12-week trial period
  Time (in terms of minutes and seconds) spent on playing tablet-based interactive games will be recorded by the game system and provided by the supplier.
The usability and acceptability of the tablet-based interactive games | At the end of the 12-week cognitive training program
  Participants and program facilitators or the next of kin of participants will complete thirteen items indicating the usability and acceptability of the tablet-based interactive games on a 5-point Likert scale (i.e. 1 indicating strongly disagree and 5 indicating strongly agree). The minimum and maximum values of the scale are 13 and 65 respectively, with higher score indicating higher usability and acceptability of games.
Change of neuropsychiatric symptoms before and after using the tablet-based interactive games | Baseline and at the end of 12-week trial period
  Change of neuropsychiatric symptoms of using the tablet-based interactive games for 12 weeks will be measured by Neuropsychiatric Inventory Questionnaire (NPI-Q). Program facilitators will complete twelve items. The range of the severity scale is 12 to 36, with higher score indicating more severe neuropsychiatric symptoms. The range of the caregiver distress scale is 0 to 60, with higher score indicating higher caregiver distress.
Change of upper-body flexibility before and after using the tablet-based interactive games | Baseline and at the end of 12-week trial period
  Change of upper-body flexibility before and after using the tablet-based interactive games will be assessed by HKU research staff who is blinded to the group allocation. The assessments of upper-body flexibility measured by Functional Reach Test. The distance in unit of centimeter of arm reach will be recorded.
Change of physical side effects before and after using digital device | Baseline and at the end of 12-week trial period
  Change of physical side effects of using digital device for 12 weeks will be measured by four items on 1. sleepless/restless sleep patterns, 2. red eyes/eye irritation/ dryness eyes, 3. shoulder or neck pain/sore muscle, and 4. retinal disease/eye pain, with 0 indicating no symptom and 2 indicating always having symptom. The minimum and maximum values of the scale are 0 and 8 respectively, with higher score indicating more physical side effects of using digital devices.
Qualitative measures: The perceived benefits and feasibility of the cognitive training program and tablet-based interactive games of participants | At the end of 12-week trial period
  A total of 2-3 participants who can communicate from each test site will be invited to participate in the qualitative interview. The contents include:
  1. What do you think about the tablet-based interactive games?
  2. What do you think about the cognitive training program?
  3. Do you want to continue to play the tablet-based interactive games in the future?
  4. Do you want to join if service unit arranges similar cognitive training program?
Qualitative measures: The perceived benefits and feasibility of the cognitive training program and tablet-based interactive games of program facilitators | At the end of 12-week trial period
  All program facilitators will be invited to participate in the qualitative interview. The contents include:
  1. What do you think about the local elements of cognitive game?
  2. Were the participants willing to play the cognitive games?
  3. Was there any improvement on cognitive functioning after the intervention program?
  4. Is it safe to play game?
  5. Is it easy to play game?
  6. Was there any abnormal situation during the trial period? Was the problem solved?
  7. Do you think the cognitive game can help on the cognitive training?
  8. What was the reaction of participants?
  9. What were your concern before playing games?
  10. Did the cognitive game fulfill your expectation?
  11. On the whole, are you satisfied with the games?
  12. To what extent, do you want the service users to continue to play the games?
  13. Do you think the time and number of scheduled training sessions was opportune?
  14. Would you recommend the games to others?
Change of the activities in daily living of person with intellectual disability before and after using the tablet-based interactive games | Baseline and at the end of 12-week trial period
  Change of the activities in daily living of all participants in rehabilitation setting will be assessed by program facilitators of the study sites. Total ten items on the Barthel Index will be completed at the baseline and the end of 12-week trial period. The minimum and maximum scores are 0 and 100 respectively, with lower score indicating higher level of dependence.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (5):
- Hong Kong (5):
  - Haven of Hope Day Care cum Rehabilitation Centre for Elderly (Hong Kong West/ Hong Kong East), Hong Kong
  - Haven of Hope Nursing Home, Hong Kong
  - Haven of Hope Rehabilitation Services for Disabled, Hong Kong
  - Haven of Hope Sister Annie Skau Holistic Care Centre, Hong Kong
  - Haven of Hope Woo Ping Care & Attention Home, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Background] Chiu HFK, Zhong BL, Leung T, Li SW, Chow P, Tsoh J, Yan C, Xiang YT, Wong M. Development and validation of a new cognitive screening test: The Hong Kong Brief Cognitive Test (HKBC). Int J Geriatr Psychiatry. 2018 Jul;33(7):994-999. doi: 10.1002/gps.4883. Epub 2018 Apr 11. PMID 29642275
- [Background] Katz-Leurer M, Fisher I, Neeb M, Schwartz I, Carmeli E. Reliability and validity of the modified functional reach test at the sub-acute stage post-stroke. Disabil Rehabil. 2009;31(3):243-8. doi: 10.1080/09638280801927830. PMID 18608433
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Tyrer SP, Wigham A, Cicchetti D, Margallo-Lana M, Moore PB, Reid BE. Comparison of short and long versions of the Prudhoe Cognitive Function Test and the K-BIT in participants with intellectual impairment. J Autism Dev Disord. 2010 Aug;40(8):1000-5. doi: 10.1007/s10803-010-0949-3. PMID 20143147
- See also: Human Benchmark (2023, Jan 26). Reaction Time Test. Human Benchmark. — https://humanbenchmark.com/tests/reactiontime